CLINICAL TRIAL: NCT00647309
Title: Correlation Between Troponin Level and Rehabilitation Outcome in Elderly Patient With Hip Fracture
Brief Title: Troponin Elevation in the Elderly Patient With Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Marina Arad, md, Sheba Medical Center
Other Study IDs: SHEBA-08-5096-MA-CTIL
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Elevated troponin is powerful and independent adverse prognostic marker in patient with ACS. However, non specific (non cardiac) troponin elevation is a common finding among hospitalized patients and worse prognosis too.

The aim of this study is examine the prevalence of incidental cardiac troponin rise in a group of patient aged 65 and over admitted to geriatric department with hip fracture, and influence of troponin elevation on outcomes like ACS, death, motor and cognitive function.

DETAILED DESCRIPTION:
data collection will include epidemiological data (age, gender, living arrangement, basic functional status, fracture date, surgery date, surgery type, length of stay) as well as previous comorbidities. in addition, routine blood tests and baseline ECG will be recorded.

troponin levels will be studied within 24 hours from admission, and 24 hours following surgery. in case of elevated troponin levels, ECG will be repeated, and echocardiography together with a cardiologist evaluation will be carried out.

data regarding in-hospital complications, motor and cognitive function (by FIM scale) and lab will be recorded. after discharge. followup will be recorded every 3 months, up to 1 year period, recoding the above mentioned data.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over with hip fracture

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 years and over with hip fracture
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
all cause mortality, motor and cognitive function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marina Arad, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Geriatric Rehabilitation dept, Ramat Gan, Israel